CLINICAL TRIAL: NCT02169453
Title: Pharmacokinetic-pharmacodynamic Interaction Between Each of Three Different Single Doses of BIA 9-1067 and a Single-dose of Controlled-release 100/25 mg Levodopa/Carbidopa: a Double-blind, Randomized, Four-way Crossover, Placebo-controlled Study in Healthy Male Subjects
Brief Title: Pharmacokinetic-pharmacodynamic Interaction Between Each of Three Different Single Doses of BIA 9-1067 and a Single-dose of Controlled-release 100/25 mg Levodopa/Carbidopa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-110
Record Dates: First submitted 2012-01-20; First posted 2014-06-23 (Estimated); Results first posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease (PD); BIA 9-1067; Opicapone
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Period 1: BIA 9-1067 25 mg Period 2: BIA 9-1067 50 mg Period 3: BIA 9-1067 100 mg Period 4: Placebo
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Sinemet® CR 100/25 (Single-dose of controlled-release levodopa/carbidopa 100/25 mg: 1 tablet of Sinemet® CR 100/25.)
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Sinemet® CR 100/25
- Group 2 (Experimental): Period 1: BIA 9-1067 50 mg Period 2: BIA 9-1067 100 mg Period 3: Placebo Period 4: BIA 9-1067 25 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Sinemet® CR 100/25 (Single-dose of controlled-release levodopa/carbidopa 100/25 mg: 1 tablet of Sinemet® CR 100/25.)
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Sinemet® CR 100/25
- Group 3 (Experimental): Period 1: BIA 9-1067 100 mg Period 2: Placebo Period 3: BIA 9-1067 25 mg Period 4: BIA 9-1067 50 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Sinemet® CR 100/25 (Single-dose of controlled-release levodopa/carbidopa 100/25 mg: 1 tablet of Sinemet® CR 100/25.)
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Sinemet® CR 100/25
- Group 4 (Experimental): Period 1: Placebo Period 2: BIA 9-1067 25 mg Period 3: BIA 9-1067 50 mg Period 4: BIA 9-1067 100 mg
  Subjects were to attend four treatment periods and were to receive a different dose of BIA 9-1067 (25 mg, 50 mg and 100 mg) or placebo during each of these treatment periods.
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Sinemet® CR 100/25

INTERVENTIONS:
Drug: BIA 9-1067 — OPC, Opicapone
  Other Names: OPC, Opicapone
Drug: Placebo — PLC, Placebo
  Other Names: PLC, Placebo
Drug: Sinemet® CR 100/25 — Controlled-release levodopa/carbidopa 100/25 mg

SUMMARY:
To investigate the effect of three single oral doses of BIA 9-1067 (25 mg, 50 mg and 100 mg) on the levodopa pharmacokinetics when administered in combination with a single-dose of controlled-release levodopa/carbidopa 100/25 mg (Sinemet® CR 100/25)

DETAILED DESCRIPTION:
Single centre, double-blind, randomized, placebo-controlled, crossover study with four consecutive single-dose treatment periods. The washout period between doses was to be at least 14 days. On each treatment period, after completion of pre-dose assessments, BIA 9-1067/Placebo was to be administered concomitantly with the dose of Sinemet® CR 100/25; post-dose assessments were to be completed and subjects were to be discharged 72 h post-dose. Subjects were to attend four treatment periods and were to receive a different dose of BIA 9-1067 (25 mg, 50 mg and 100 mg) or placebo during each of these treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the entire study period and willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer prior to participation in the study.
* Male volunteers.
* Volunteers of at least 18 years of age but not older than 45 years.
* Volunteers with body mass index (BMI) greater than or equal to 19 and below 30 kg/m2.
* Volunteers who were non- or ex-smokers. An ex-smoker is defined as someone who completely stopped smoking for at least 12 months before day 1 of this study.
* Volunteers who were healthy as determined by pre-study (at screening) medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Volunteers who had clinical laboratory test results judged clinically acceptable (within the laboratory's stated normal range; if not within this range, they must had been without any clinical significance) at screening and admission to first treatment period.
* Volunteers who had negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C antibodies (HCV Ab), and Human immunodeficiency viruses -1 and -2 antibodies (HIV-1 and HIV-2 Ab) at screening.
* Volunteers who had negative screen of ethyl alcohol and drugs of abuse at screening.
* Due to unknown risks and potential harm to the unborn fetus, sexually active men must have agreed to use a medically acceptable form of contraception throughout the study.

Exclusion Criteria:

* Volunteers who did not conform to the above inclusion criteria, or in case of
* Volunteers who had a clinically relevant surgical history.
* Volunteers who had a clinically relevant family history.
* Volunteers who had a history of relevant atopy.
* Volunteers who had a significant infection or known inflammatory process at screening or first admission.
* Volunteers who had acute gastrointestinal symptoms at the time of screening or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Volunteers who were vegetarians, vegans or have medical dietary restrictions.
* Volunteers who could not communicate reliably with the investigator.
* Volunteers who were unlikely to co-operate with the requirements of the study.
* Significant history of hypersensitivity to BIA 9-1067, tolcapone, entacapone, levodopa, carbidopa or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability.
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, lymphatic, musculoskeletal, genitourinary, endocrine, immunologic, dermatologic or connective tissue disease.
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases.
* Presence of significant heart disease or disorder according to ECG.
* Presence of suspicious undiagnosed skin lesions or a history of melanoma.
* Previous history of Neuroleptic Malignant Syndrome (NMS) and/or nontraumatic rhabdomyolysis.
* Presence or history of significant glaucoma.
* Used of prescription medications including monoamine oxidase (MAO) inhibitors within 28 days before day 1 of the study.
* Used of over-the-counter (OTC) products within 7 days before day 1 of the study.
* Maintenance therapy with any drug, or significant history of drug dependency (drug abuse) or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
* Any clinically significant illness in the previous 28 days before day 1 of this study.
* Used of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin and rifampicin), in the previous 28 days before day 1 of this study.
* Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study.
* Poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician.
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study.
* Positive urine screening of ethyl alcohol or drugs of abuse at admission to any treatment period.
* Any history of tuberculosis and/or prophylaxis for tuberculosis.
* Positive results to HIV, HBsAg or anti-HCV tests.
* Participation in any previous clinical study with BIA 9-1067 within 84 days before day 1 of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Algorithme Pharma Inc, Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Period 1: BIA 9-1067 25 mg Period 2: BIA 9-1067 50 mg Period 3: BIA 9-1067 100 mg Period 4: Placebo
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Sinemet® CR 100/25 (Single-dose of controlled-release levodopa/carbidopa 100/25 mg: 1 tablet of Sinemet® CR 100/25.)
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Sinemet® CR 100/25: Controlled-release levodopa/carbidopa 100/25 mg
- Group 2: Period 1: BIA 9-1067 50 mg Period 2: BIA 9-1067 100 mg Period 3: Placebo Period 4: BIA 9-1067 25 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Sinemet® CR 100/25 (Single-dose of controlled-release levodopa/carbidopa 100/25 mg: 1 tablet of Sinemet® CR 100/25.)
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Sinemet® CR 100/25: Controlled-release levodopa/carbidopa 100/25 mg
- Group 3: Period 1: BIA 9-1067 100 mg Period 2: Placebo Period 3: BIA 9-1067 25 mg Period 4: BIA 9-1067 50 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Sinemet® CR 100/25 (Single-dose of controlled-release levodopa/carbidopa 100/25 mg: 1 tablet of Sinemet® CR 100/25.)
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Sinemet® CR 100/25: Controlled-release levodopa/carbidopa 100/25 mg
- Group 4: Period 1: Placebo Period 2: BIA 9-1067 25 mg Period 3: BIA 9-1067 50 mg Period 4: BIA 9-1067 100 mg
  Subjects were to attend four treatment periods and were to receive a different dose of BIA 9-1067 (25 mg, 50 mg and 100 mg) or placebo during each of these treatment periods.
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Sinemet® CR 100/25: Controlled-release levodopa/carbidopa 100/25 mg
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 3 | 3 | 3 | 3
25 mg BIA 9-1067 | 3 | 3 | 3 | 3
50 mg BIA 9-1067 | 3 | 3 | 2 | 3
100 mg BIA 9-1067 | 3 | 3 | 3 | 3
Placebo | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Cmax - Maximum observed plasma concentration of levodopa
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 25 mg: BIA 9-1067 25 mg OPC Opicapone
- BIA 9-1067 50 mg: BIA 9-1067 50 mg OPC Opicapone
- BIA 9-1067 100 mg: BIA 9-1067 100 mg OPC Opicapone
- Placebo: Placebo, PLC
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 12 | 12
ng/mL | 716 (201.9) | 673 (269.9) | 570 (136.2) | 554 (220.5)

2. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve to Last Measurable Time Point
Description: AUC0-t - Area under the plasma concentration-time curve to last measurable time point for levodopa
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 12 | 12
ng.h/mL | 1886 (396.1) | 1997 (389.4) | 2059 (372.7) | 1575 (521.3)

3. Primary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve Extrapolated to Infinity
Description: AUC0-∞ - Area under the plasma concentration-time curve extrapolated to infinity for levodopa
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 12 | 12
ng.h/mL | 1986 (395.2) | 2144 (437.4) | 2215 (381.0) | 1677 (541.7)

4. Primary Outcome: Emax - Maximum Inhibition of COMT Activity
Description: Emax - Maximum inhibition of Catechol-O-Methyltransferase (COMT) activity
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose
Measure: Mean (Standard Deviation); unit: pmol/mg Hb/h
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 12 | 12
pmol/mg Hb/h | 16.5 (10.8) | 7.44 (7.42) | 3.16 (4.97) | 39.3 (16.0)

5. Primary Outcome: tEmax - Time of Occurrence of Emax
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 12 | 12
hours | 4.92 (2.71) | 3.59 (1.95) | 2.33 (0.985) | 7.17 (8.95)

6. Primary Outcome: AUEC0-24 - Area Under the Effect-time Curve From t=0h to t=24h
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose
Measure: Mean (Standard Deviation); unit: pmol/mg Hb/h.h
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 12 | 11 | 12 | 12
pmol/mg Hb/h.h | 621 (300) | 427 (214) | 363 (201) | 1144 (445)

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 4/11 | 4/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 25 mg (N=12) | BIA 9-1067 50 mg (N=11) | BIA 9-1067 100 mg (N=12) | Placebo (N=12)
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Application site erythema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 2
Feeling hot (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram PR interval (Investigations) | 0 | 0 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 2 | 0 | 3
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1
Impatience (Psychiatric disorders) | 1 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 1
Terminal dribbling (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other